CLINICAL TRIAL: NCT07190846
Title: Diastolic Dysfunction in the Pregnant Woman With Preeclampsia
Brief Title: Diastolic Dysfunction 2025
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, Associate Professor of Anesthesiology and Critical Care, Principal Investigator, University Tunis El Manar
Other Study IDs: 05/2025
Record Dates: First submitted 2025-09-01; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia; Severe Preeclampsia
Keywords: Diastolic dysfunction; Echocardiography; Maternal heart function; Left ventricular relaxation; Pregnancy hypertension; Cardio-obstetrics; Maternal cardiovascular risk
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preeclampsia Group: Pregnant women in the third trimester diagnosed with preeclampsia (mostly severe forms), aged 18-45 years, without pre-existing cardiovascular disease or other exclusion criteria.
  Interventions: Other: No Intervention (Observational Echocardiographic Evaluation)
- Control Group: Normotensive pregnant women in the third trimester, aged 18-45 years, without cardiovascular disease or other exclusion criteria.
  Interventions: Other: No Intervention (Observational Echocardiographic Evaluation)

INTERVENTIONS:
Other: No Intervention (Observational Echocardiographic Evaluation) — This is an observational study. No therapeutic intervention is administered. Participants undergo standard echocardiographic assessment of left ventricular diastolic function during pregnancy.

SUMMARY:
This is a prospective observational study conducted at the Maternity and Neonatology Center of Tunis to evaluate cardiac diastolic function in women with preeclampsia compared with normotensive pregnant women. A total of 80 pregnant women in the third trimester were enrolled, including 40 with preeclampsia (mostly severe forms) and 40 healthy controls. All participants underwent standardized transthoracic echocardiography to assess left ventricular diastolic function according to the 2016 ASE/EACVI recommendations.

DETAILED DESCRIPTION:
Preeclampsia is a major hypertensive disorder of pregnancy associated with increased maternal morbidity and mortality, as well as long-term cardiovascular risk. Cardiac remodeling in this context is characterized by increased vascular stiffness and concentric left ventricular hypertrophy, which may lead to subclinical diastolic dysfunction despite preserved systolic function.

This prospective observational study was designed to evaluate left ventricular diastolic function in women with preeclampsia compared to normotensive pregnant women. Eighty participants in the third trimester of pregnancy were included: 40 diagnosed with preeclampsia (mainly severe forms) and 40 normotensive controls. Women with pre-existing cardiovascular disease, diabetes, renal impairment, or multiple pregnancies were excluded.

All participants underwent standardized echocardiographic evaluation in accordance with the 2016 recommendations of the American Society of Echocardiography (ASE) and the European Association of Cardiovascular Imaging (EACVI). Diastolic function was assessed based on transmitral Doppler indices (E and A waves, E/A ratio), tissue Doppler imaging (septal and lateral e' velocities), E/e' ratio, left atrial volume index, and tricuspid regurgitation velocity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-45 years
* Third trimester of pregnancy
* Group A: women diagnosed with preeclampsia according to international criteria (blood pressure ≥ 140/90 mmHg after 20 weeks with proteinuria or signs of severity)
* Group B (controls): normotensive pregnant women without proteinuria or cardiovascular disease
* Signed informed consent

Exclusion Criteria:

* Known pre-existing cardiovascular disease (structural heart disease, heart failure, chronic hypertension complicated)
* Left ventricular ejection fraction < 45%
* Pre-gestational diabetes
* Chronic kidney disease
* Multiple pregnancy
* Other severe comorbidities that could affect cardiac function independently of preeclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women in the third trimester recruited at the Center of Maternity and Neonatology of Tunis, including 40 with preeclampsia (mainly severe forms) and 40 normotensive controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Left Ventricular Diastolic Dysfunction in Preeclamptic Women | At baseline, during third-trimester pregnancy hospital evaluation.
  Echocardiographic assessment of diastolic function according to ASE/EACVI 2016 criteria, including parameters E, A, E/A ratio, septal and lateral e' velocities, E/e' ratio, left atrial volume index, and tricuspid regurgitation velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Ben marzouk sofiene, Principal Investigator — Maternity and Neonatology Center of Tunis
Locations (1):
- Maternity and Neonatology Center of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet decided whether individual participant data (IPD) from this study will be shared. Decisions regarding data sharing will depend on future institutional policies, ethical considerations, and requests from qualified researchers.

REFERENCES:
- [Result] Soma-Pillay P, Louw MC, Adeyemo AO, Makin J, Pattinson RC. Cardiac diastolic function after recovery from pre-eclampsia. Cardiovasc J Afr. 2018 Jan/Feb 23;29(1):26-31. doi: 10.5830/CVJA-2017-031. Epub 2017 Aug 31. PMID 28906533
- [Result] Guirguis GF, Aziz MM, Boccia Liang C, Williams SF, Apuzzio JJ, Bilinski R, Mornan AJ, Shah LP. Is preeclampsia an independent predictor of diastolic dysfunction? A retrospective cohort study. Pregnancy Hypertens. 2015 Oct;5(4):359-61. doi: 10.1016/j.preghy.2015.10.001. Epub 2015 Oct 9. PMID 26597754
- [Result] Vaught AJ, Kovell LC, Szymanski LM, Mayer SA, Seifert SM, Vaidya D, Murphy JD, Argani C, O'Kelly A, York S, Ouyang P, Mukherjee M, Zakaria S. Acute Cardiac Effects of Severe Pre-Eclampsia. J Am Coll Cardiol. 2018 Jul 3;72(1):1-11. doi: 10.1016/j.jacc.2018.04.048. PMID 29957219
- [Result] Melchiorre K, Sutherland GR, Baltabaeva A, Liberati M, Thilaganathan B. Maternal cardiac dysfunction and remodeling in women with preeclampsia at term. Hypertension. 2011 Jan;57(1):85-93. doi: 10.1161/HYPERTENSIONAHA.110.162321. Epub 2010 Nov 22. PMID 21098311
- [Result] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT07190846/Prot_SAP_000.pdf